CLINICAL TRIAL: NCT06051175
Title: Effect of Food Sensorial Perception on Brain Activity, Cardiovascular Activity, Facial Mimicry and Electrodermal Activity
Brief Title: Study of the Neurophysiological Response to Foodstuffs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 1226Neurophy
Record Dates: First submitted 2023-09-07; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Healthy Nutrition
Keywords: sensory perception; physiological response; neurophysiological response; basic flavour
MeSH Terms: interventions — Candy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sensory attributes perception - bitter taste (Experimental): During the experiment individuals will be exposed to caffeine solution, identifying the sensory attributes and basic flavours. Between the tastings of the different foodstuffs, neutralisation phases will occur, where participants will receive a neutral food stimulus. The judgement will be self-reported by the participants after contact with the food.
  While the study is taking place, physiological and neurophysiological data will be collected from participants: brain activity (EEG); cardiac activity (ECG); electrodermal activity (galvanic skin response); and facial mimicry via video analysis and eye tracking. These data will be analysed using physiological data analysis software. All participant data will be recorded using coding, ensuring anonymity and confidentiality.
  Interventions: Other: Bitter taste perception
- Sensory attributes perception - salty taste (Experimental): Individuals will be exposed to sodium chloride solution, identifying the sensory attributes and basic flavours. Between the tastings of the different foodstuffs, neutralisation phases will occur, where participants will receive a neutral food stimulus. The judgement will be self-reported by the participants after contact with the food.
  While the study is taking place, physiological and neurophysiological data will be collected from participants: brain activity (EEG); cardiac activity (ECG); electrodermal activity (galvanic skin response); and facial mimicry via video analysis and eye tracking. These data will be analysed using physiological data analysis software. All participant data will be recorded using coding, ensuring anonymity and confidentiality.
  Interventions: Other: Salty taste perception
- Sensory attributes perception - sweet taste (Experimental): Individuals will be exposed to sucrose solution, identifying the sensory attributes and basic flavours. Between the tastings of the different foodstuffs, neutralisation phases will occur, where participants will receive a neutral food stimulus. The judgement will be self-reported by the participants after contact with the food.
  While the study is taking place, physiological and neurophysiological data will be collected from participants: brain activity (EEG); cardiac activity (ECG); electrodermal activity (galvanic skin response); and facial mimicry via video analysis and eye tracking. These data will be analysed using physiological data analysis software. All participant data will be recorded using coding, ensuring anonymity and confidentiality.
  Interventions: Other: Sweet taste perception
- Sensory attributes perception - acid taste (Experimental): Individuals will be exposed to citric acid solution, identifying the sensory attributes and basic flavours. Between the tastings of the different foodstuffs, neutralisation phases will occur, where participants will receive a neutral food stimulus. The judgement will be self-reported by the participants after contact with the food.
  While the study is taking place, physiological and neurophysiological data will be collected from participants: brain activity (EEG); cardiac activity (ECG); electrodermal activity (galvanic skin response); and facial mimicry via video analysis and eye tracking. These data will be analysed using physiological data analysis software. All participant data will be recorded using coding, ensuring anonymity and confidentiality.
  Interventions: Other: Acid taste perception
- Sensory attributes perception - umami taste (Experimental): Individuals will be exposed to sodium glutamate monohydrate solution, identifying the sensory attributes and basic flavours. Between the tastings of the different foodstuffs, neutralisation phases will occur, where participants will receive a neutral food stimulus. The judgement will be self-reported by the participants after contact with the food.
  While the study is taking place, physiological and neurophysiological data will be collected from participants: brain activity (EEG); cardiac activity (ECG); electrodermal activity (galvanic skin response); and facial mimicry via video analysis and eye tracking. These data will be analysed using physiological data analysis software. All participant data will be recorded using coding, ensuring anonymity and confidentiality.
  Interventions: Other: Umami taste perception

INTERVENTIONS:
Other: Bitter taste perception — Participants will perform a bitter taste perception analysis. During the analysis of sensory attributes, participants will pass the solutions through the various regions of the tongue, and at the end, throw the contents away, not ingesting the solution. Between analyzing the various solutions, participants will rinse their mouth with water.
  Simultaneously with the analysis of sensory attributes, each participant will be subjected to an assessment of brain activity and physiological activity through the following non-invasive methods: electroencephalography technique; electrocardiography technique; monitoring cardiac electrical activity; facial mimicry activity via video analysis and eye tracking; and electrodermal activity using galvanic skin response.
  Arms: Sensory attributes perception - bitter taste
Other: Salty taste perception — Participants will perform a salty taste perception analysis. During the analysis of sensory attributes, participants will pass the solutions through the various regions of the tongue, and at the end, throw the contents away, not ingesting the solution. Between analyzing the various solutions, participants will rinse their mouth with water.
  Simultaneously with the analysis of sensory attributes, each participant will be subjected to an assessment of brain activity and physiological activity through the following non-invasive methods: electroencephalography technique; electrocardiography technique; monitoring cardiac electrical activity; facial mimicry activity via video analysis and eye tracking; and electrodermal activity using galvanic skin response.
  Arms: Sensory attributes perception - salty taste
Other: Sweet taste perception — Participants will perform a sweet taste perception analysis. During the analysis of sensory attributes, participants will pass the solutions through the various regions of the tongue, and at the end, throw the contents away, not ingesting the solution. Between analyzing the various solutions, participants will rinse their mouth with water.
  Simultaneously with the analysis of sensory attributes, each participant will be subjected to an assessment of brain activity and physiological activity through the following non-invasive methods: electroencephalography technique; electrocardiography technique; monitoring cardiac electrical activity; facial mimicry activity via video analysis and eye tracking; and electrodermal activity using galvanic skin response.
  Arms: Sensory attributes perception - sweet taste
Other: Acid taste perception — Participants will perform a acid taste perception analysis. During the analysis of sensory attributes, participants will pass the solutions through the various regions of the tongue, and at the end, throw the contents away, not ingesting the solution. Between analyzing the various solutions, participants will rinse their mouth with water.
  Simultaneously with the analysis of sensory attributes, each participant will be subjected to an assessment of brain activity and physiological activity through the following non-invasive methods: electroencephalography technique; electrocardiography technique; monitoring cardiac electrical activity; facial mimicry activity via video analysis and eye tracking; and electrodermal activity using galvanic skin response.
  Arms: Sensory attributes perception - acid taste
Other: Umami taste perception — Participants will perform a umami taste perception analysis. During the analysis of sensory attributes, participants will pass the solutions through the various regions of the tongue, and at the end, throw the contents away, not ingesting the solution. Between analyzing the various solutions, participants will rinse their mouth with water.
  Simultaneously with the analysis of sensory attributes, each participant will be subjected to an assessment of brain activity and physiological activity through the following non-invasive methods: electroencephalography technique; electrocardiography technique; monitoring cardiac electrical activity; facial mimicry activity via video analysis and eye tracking; and electrodermal activity using galvanic skin response.
  Arms: Sensory attributes perception - umami taste

SUMMARY:
The goal of this clinical trial is to investigate the effect of perception of sensory attributes of different foodstuffs on physiological and neurophysiological response in health adults. The main aims are:

* To evaluate the effect of sensory perception of foodstuffs on brain activity using EEG technique;
* To evaluate the effect of food sensory perception on cardiovascular activity using EGG;
* To evaluate the effect of food sensory perception on facial mimicry via video analysis and eye tracking;
* To evaluate the effect of food sensory perception on electrodermal activity using galvanic skin response.

Participants will perform a sensory attribute perception analysis of 5 different solutions representing basic flavours. During the analysis of sensory attributes, participants will pass the solutions through the various regions of the tongue, and at the end, throw the contents away, not ingesting the solution. Between analyzing the various solutions, participants will rinse their mouth with water.

Simultaneously with the analysis of sensory attributes, each participant will be subjected to an assessment of brain activity and physiological activity through the following non-invasive methods: electroencephalography technique; electrocardiography technique; monitoring cardiac electrical activity; facial mimicry activity via video analysis and eye tracking; and electrodermal activity using galvanic skin response.

DETAILED DESCRIPTION:
Participation in the Study of the neurophysiological response to foodstuffs in university students with the aim of investigating the effect of the perception of the sensory attributes of different foodstuffs on the physiological and neurophysiological response of healthy university students, which consists of the following participation: Completion of a survey with the aim of finding out the participant's family history in terms of pathologies and/or allergies/intolerances, gender, age, medication, smoking habits and lifestyles, anthropometric data.

Participants will carry out an analysis of the perception of sensory attributes of 5 different solutions representing basic flavours. During the analysis of sensory attributes, the participants will have to pass the solutions over the various regions of the tongue, and at the end, throw the contents away, not ingesting the solution. Between analysing the various solutions, participants will rinse their mouths out with water.

Simultaneously with the analysis of sensory attributes, each participant will undergo an assessment of brain activity and physiological activity using the following non-invasive methods: Electroencephalography technique, which consists of monitoring brain electrical activity using a cap with electrodes on the head. The electrocardiography technique, which consists of monitoring cardiac electrical activity by placing 3 electrodes on the forearm. Facial mimicry via video analysis and eye tracking, which consists of monitoring facial mimicry by recording test videos for each participant. The participant will be recorded throughout the experiment. Electrodermal activity using the galvanic response of the skin, where the participant will place their index finger and middle finger on a sensor for analysis. The evaluation of brain activity, which includes all the techniques described above, lasts a maximum of one hour.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* agree to take part in the study
* aged between 18 and 25

Exclusion Criteria:

* Participants with cardiovascular, neurological or psychiatric conditions
* Participants with food allergies or intolerances
* Participants with disability that does not allow them to fully utilise their sense of taste (ageusia) and smell (anosmia).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
The mean value of electroencephalography signal components at different flavours | During the intervention
  The mean value of electroencephalography (EEG) signal components delta (1-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), low-beta (12-20 Hz), high-beta (20-30 Hz) and gamma (30-45 Hz) (in decibel) will be measure by the EEG raw signals recorded by a 64-channel EEG device for each flavour
Mean score of valence, arousal, dominance in the Self Assessment Manikin System for each flavour | Immediately after the intervention
  The characterization of the flavour is performed using a 9-point scale for quantifying valence (pleasant/unpleasant), arousal (exciting/calming) and dominance (overwhelming/subtle)
The mean value of heart rate and heart rate variability computed from the electrocardiography raw signal at different flavours | During the intervention
  The mean value of heart rate (in beats per minute), the heart rate variability (in milliseconds) and will be measure bt the electrocardiography (ECG) raw signal recorded by an ECG device for each flavour
The left and right pupil dilatation at different flavours | During the intervention
  The left and right pupil dilatation will be extracted from the eye tracker device
The electrodermal activity values at different flavours | During the intervention
  The electrodermal activity, namely the skin conductance response and skin conductance level (in microSiemens) will be directly measure by Galvanic skin response device
Facial expressions induced by different flavours | During the intervention
  The facial expressions (in action units) will be visually measured on the videos that were acquired using a camera

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Universitário Egas Moniz, Almada, Monte de Caparica, Portugal